Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

NCT #: NCT04506307

# Noninvasive Fat Reduction with the CoolSculpting System

## **Investigational Plan**

| Sponsor | ZELTIQ Aesthetics, Inc., An Allergan Affiliate<br>4410 Rosewood Dr.<br>Pleasanton, CA 94588 |
|---|---|
| Protocol Number: | ZA20-001 |
| Protocol Version: | 04 |
| Protocol Date: | 19 September 2022 |
| Product (s) | CoolSculpting System |
| Sponsor Contact: | PH: Email: |

Part Number: CS-305578 Revision: 04  Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

| Part Number: CS-305578 | Revision: 04 |
|---|---|
| Title: Noninvasive Fat Redu | ction with the CoolSculpting System |



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

| Part Number: CS-305578 | Revision: 04 | |
|---|---|---|
| Title: Noninvasive Fat Reduction | on with the CoolSculpting Sy | /stem |
| INIVESTICATOR SIGNATUR | EDACE | |
| INVESTIGATOR SIGNATUR | E PAGE | |
| For protocol number ZA20-001 | | |
| I agree to: | | |
| 8 | | |
| <u> </u> | is study diligently and in stri | <u> </u> |
| protocol, GCP, and all app | olicable laws and regulations. | • |
| Maintain all information s | upplied by the Sponsor, ZEL | TIO Aesthetics, an |
| | dence and, when this information | = |
| | d (IRB) or Ethics Committee | · /· |
| it will be submitted with a | designation that the material | l is confidential. |
| I have read this protocol in its en | ntirety and I agree to all aspe | ects. |
| Investigator printed name | Signature | Date |
| Investigator printed name | Signature | Date |
| = = = | = | |

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### **RETURN PAGE TO SPONSOR**

Part Number: CS-305578 Revision: 04

Title: Noninvasive Fat Reduction with the CoolSculpting System

## **Table of Contents**


| 1. | Pro | toc | ol Summary | 9 |
|---|---|---|---|---|
| 2. | Inti | rodu | uction | . 11 |
| | 2.1. | Ba | ckground | 11 |
| | 2.2. | Re | gulatory Status | 12 |
| | 2.3. | | | 13 |
| 3. | Dev | vice | Description | . 13 |
| 4. | Stu | dy C | Objectives | . 14 |
| 5. | Inv | esti | gational Plan | . 14 |
| | 5.1. | Stı | ıdy Design | 14 |
| | 5.2. | Inv | vestigator Qualifications | 14 |
| | 5.3. | Stı | ıdy Population | 15 |
| | 5.3. | 1. | Target Patient Population | 15 |
| | 5.3. | 2. | Subject Eligibility | 15 |
| | 5.3. | 3. | Vulnerable Populations | 16 |
| 6. | Stu | dy ( | Conduct and Procedures | . 16 |
| | 6.1. | Re | cruitment | 16 |
| | 6.2. | Inf | formed Consent | 16 |
| | 6.3. | Sci | reening Procedures | 17 |
| | 6.4. | | | 18 |
| | 6.5. | | | 18 |
| | 6.6. | Tr | eatment Procedures | 19 |
| | 6.6. | 1. | Treatment Visit #1; Required; Day 0 | 19 |
| | 6.6. | 2. | Treatment Visit #2; Required; 6 Weeks (± 1 week) | 20 |
| | 6.7. | Fo | llow-up Procedures | 21 |
| | 6.7. | 1. | One-Week Phone Follow-Up (post-each treatment); Required: 7 Days (± 3 | |
| | day | s) | 21 | |
| | 6.7. | 2. | | 21 |
| | 6.7. | 3. | Twelve-Week Final Follow-up; Required (Day 90 +/- 14 days post-treatmer 22 | nt) |
| | 6.7. | 4. | Optional Follow-Up Evaluations (up to 2 within study period) | 22 |
| | 6.8. | | | 24 |
| | 6.8. | 1. | | 24 |
| | 6.8. | 2. | | 24 |

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04  Title: Noninvasive Fat Reduction with the CoolSculpting System

| 6.8.3. | | 25 |
|---|---|---|
| 6.8.4. | | 25 |
| 6.8.5. | | 26 |
| 7. Statist | ical Methodology and Analyses | 26 |
| 7.1. <b>P</b> 1 | rimary Endpoints | 26 |
| 7.2. St | atistical Methods: Overall Plan | 26 |
| 7.3. <b>A</b> | nalysis Cohorts | 26 |
| 7.3.1. | Safety Cohort | 26 |
| 7.3.2. | Effectiveness Cohorts | 26 |
| 7.3.3. | Endpoint Analysis | 27 |
| 7.3.4. | Missing Data Handling: | 27 |
| 7.3.5. | Data Pooling: | 28 |
| 7.3.6. | | 28 |
| 8. Adver | se Events | 28 |
| | dverse Device Effect (ADE) | |
| 8.1.1. | Serious Adverse Device Effect (SADE) | |
| 8.1.2. | Unanticipated Serious Adverse Device Effect (USADE) | |
| 8.1.3. | Serious Adverse Event (SAE) | |
| 8.1.4. | Time Period and Frequency for Collecting AE and SAE Information | |
| 8.1.5. | Method of Detecting AEs and SAEs | |
| 8.1.6. | Follow-up of AEs and SAEs | |
| 8.1.7. | Reportable Incidents | |
| 8.1.8. | Assessment of Severity | 32 |
| 8.1.9. | Assessment of Relatedness | 32 |
| 8.1.10. | Serious Adverse Event Reporting Procedures | 35 |
| 8.1.11. | Pregnancy | 36 |
| 9. Device | · Tracking | 36 |
| | evice Packaging and Labeling | |
| 10. Dev | ice Deficiencies and Malfunctions | 3/ |
| 11. Ethi | cal and Regulatory Considerations | |
| 11.1. | Compliance with Good Clinical Practice | 37 |
| 11.2. | Institutional Review Board (IRB) and Informed Consent | |
| 11.3. | Protocol Adherence | |
| 11.4. | Protocol Amendments | 38 |
| 12. Stud | ly Management and Quality Control | 39 |

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

| Part Number: CS-305578 | Revision: 04 |
|---|---|
| Title: Noninvasive Fat Reduc | ction with the CoolSculpting System |

| 12.1. | Study Data Collection | 39 |
|--------|-------------------------------|----|
| 12.2. | Data Management | 39 |
| 12.2. | | |
| 12.3. | Confidentiality | 39 |
| 12.4. | Quality Assurance Audits | |
| 12.5. | Investigator Responsibilities | 40 |
| 12.5. | 1. General Responsibilities | 40 |
| 12.5. | 2. Investigator Records | 41 |
| 12.5. | 3. Investigator Reports | 42 |
| 12.6. | Sponsor Responsibilities | 43 |
| 12.6. | 1. General Responsibilities: | 43 |
| 12.6. | 2. Site Monitoring | 44 |
| 12.6. | 3. Final Report | 46 |
| 12.6. | 4. Trial Registration | 46 |
| 13. Da | ata Ownership | 46 |
| 14. | | 46 |
| 15. | | 46 |
| 15.1. | | |
| 15.2. | | 47 |

| Part Number: CS-305578 | Revision: 04 |
|---|---|
| Title: Noninvasive Fat Redu | ction with the CoolSculpting System |

## 1. Protocol Summary

| Title | Noninvasive Fat Reduction with the CoolSculpting System |
|---|---|
| Design | Prospective, open-label interventional study |
| Objective/Purpose | Evaluate the safety and efficacy of multiple, simultaneous CoolSculpting cycles for the purpose of non-invasive fat reduction |
| Enrollment | Up to 60 subjects |
| Clinical Sites | Up to 6 investigational sites |
| Participant/ | Healthy adult men and women aged 22 – 65 who desire |
| Subject population | non-invasive fat reduction in the torso |
| Treatment | Upon qualification, each subject will receive 2 treatment sessions, 6 weeks apart with the CoolSculpting System. At each treatment visit, multiple simultaneous cooling cycles will be performed on areas of the torso (abdomen, flanks and/or back) identified for fat reduction using CoolSculpting System applicators. A minimum of 8 (eight) cooling cycles will be performed throughout the evaluation. Follow-up visits are scheduled at 4 weeks and 12 weeks post-final treatment; phone follow-up will occur 1 week after each treatment visit. |
| Primary Endpoint(s) | Safety endpoint: The frequency of device and procedure-related adverse events (AEs), including device-related serious adverse events (SADEs), will be summarized. Efficacy endpoint: Correct identification of pre-treatment vs. 12-week post-treatment images by at least two out of three blinded, independent reviewers. Success will be |

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

| Part Number: CS-305578 | Revision: 04 |
|---|---|
| Title: Noninvasive Fat Reduc | ction with the CoolSculpting System |

| | defined as at least 70% correct identification of the pretreatment images. |
|---|---|
| Sponsor | ZELTIQ Aesthetics, Inc., An Allergan Affiliate<br>4410 Rosewood Dr.<br>Pleasanton, CA 94588 |

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### 2. Introduction

## 2.1. Background

Fat reduction and body contouring procedures, which include invasive, minimally-invasive, and non-invasive procedures, have become increasingly popular aesthetic procedures. Patients who are obese and do not have specific fat bulges but require significant fat reduction to achieve aesthetic results are candidates for invasive and minimally-invasive procedures, such as liposuction and laser-assisted liposuction. Although effective at reducing fat, these invasive and minimally-invasive procedures involve significant patient discomfort, expense, downtime, and the risks typically associated with surgical procedures. As a result, patients who do not require significant fat reduction to achieve meaningful aesthetic results typically seek non-invasive fat reduction and body contouring procedures to avoid the pain, expense, downtime, and surgical risks associated with invasive and minimally-invasive procedures.

ZELTIQ Aesthetics has developed and commercialized a technology for cold-assisted lipolysis. The ZELTIQ CoolSculpting technology is based on the sensitivity of fat cells to cold injury in order to selectively eliminate subcutaneous fat tissue without affecting the skin or other surrounding tissues. The technology, cryolipolysis, enables a non-invasive alternative for subcutaneous fat reduction through cellular apoptosis. The ZELTIQ CoolSculpting System is cleared for use in the United States for the indication of cold-assisted lipolysis of various body areas, including the upper arm, bra fat, back fat, banana roll, thigh, abdomen, and flank in individuals with a body mass index (BMI) of 30 or less. In addition, the device is intended for cold-assisted lipolysis of the submental and submandibular areas in individuals with a BMI up to 46.2. The CoolSculpting System has been clinically proven to reduce fat bulges, allowing patients to achieve noticeable and measurable aesthetic results without the pain, expense, downtime, and risks associated with existing invasive and minimally-invasive procedures.

Clinical studies of the CoolSculpting System used on the abdomen have demonstrated the treatment to be safe and effective for the reduction of subcutaneous fat. Subjects in a recent study rated their satisfaction with the

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

CoolSculpting procedure at 73% and 89% indicated they would recommend the procedure. <sup>1</sup>

While the CoolSculpting procedure is successful in reducing subcutaneous fat in various anatomical areas, patients often desire treatment in multiple body areas (e.g. abdomen and flanks) necessitating serial treatment sessions to achieve desired results. Physician feedback suggests patients would prefer to have multiple CoolSculpting cycles performed at once in a single office visit to reduce the overall time of the procedures. ZELTIQ is exploring the simultaneous use of multiple CoolSculpting applicators to reduce overall treatment time and improve body contouring effects for multiple body areas.

Zeltiq has enhanced the CoolSculpting System to accommodate simultaneous use of two applicators. The new system, the CoolSculpting Elite System, is under investigation in this evaluation. The purpose of this trial is to further evaluate the safety and efficacy of the CoolSculpting Elite System when multiple cooling cycles are applied simultaneously to the torso for non-invasive subcutaneous fat reduction.

#### 2.2. Regulatory Status

The CoolSculpting System has been cleared in the United States for use as an aesthetic treatment to affect the appearance of the flanks (DEN090002), abdomen (K120023), thighs (K133212), arms (K162050), submental area, (K181740) submandibular area (K151179), and bra fat, back fat, and banana roll (K160259). Additionally, the System has been cleared for flexible treatment parameter ranges (K142491). FDA clearance allows treatment duration of up to 120 minutes, and at temperatures as low as -15°C.

<sup>&</sup>lt;sup>1</sup> Krueger, N., Mai, S. V., Luebberding, S., & Sadick, N. S. (2014). Cryolipolysis for noninvasive body contouring: clinical efficacy and patient satisfaction. *Clinical, cosmetic and investigational dermatology*, 7, 201.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

The device was also previously cleared for cooling as a method to minimize localized pain and thermal injury during laser and dermatological treatments under: K060407 (initial clearance), K063715 (clearance for warming and massage), K072152 (clearance for flat and belt applicators), K080118 (clearance for vacuum applicator), and K090094 (clearance for commercial device) and K193566 (clearance for updated CoolSculpting System).



## 3. Device Description

The CoolSculpting Elite System is comprised of a control unit (**Figure 1**) which houses the system controller and power source, and two detachable applicators that are used to apply the cooling and/or warming to the treatment site. The applicators use vacuum pressure to draw tissue into the cup shaped applicator. The applicator types to be used in this study are the CoolSculpting family of applicators. (**Figure 2**). Physicians will select an appropriately sized applicator for the body area(s) intended for treatment. All applicators will be used with cooling cycle parameters of a temperature of -11°C, and treatment duration of 35 minutes or 45 minutes (as appropriate by applicator type).



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



## 4. Study Objectives

The objectives of the trial are to determine the safety and effectiveness of performing multiple simultaneous cooling cycles on the torso with the CoolSculpting Elite System.

## 5. Investigational Plan

Upon qualification, each subject will receive 2 treatments sessions 6 weeks apart with the CoolSculpting Elite system. At each treatment visit, multiple simultaneous cooling cycles will be performed on areas of the torso (abdomen, flanks and/or back) identified for fat reduction using CoolSculpting System applicators. A minimum of 8 (eight) cooling cycles will be performed throughout the study. Follow-up visits are scheduled at 4 weeks after each treatment visit and 12 weeks post-final treatment; phone follow-up will occur 1 week after each treatment visit.

## 5.1. Study Design

Up to 6 sites will enroll 60 eligible subjects in this prospective, interventional, non-randomized open-label study. Enrollment and follow-up is expected to take up to five (5) months for each subject. The completion time for enrollment is anticipated to be 5 months, with the total study duration expected to be approximately 10 months.

## 5.2. Investigator Qualifications

To participate in this study, an Investigator must have an active medical license and board certification in dermatology and/or plastic surgery. The investigator must undergo training on the study device(s) prior to study initiation.

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

Site investigators must have at least one study coordinator with experience in conducting aesthetic research and with sufficient time to conduct the study.

## 5.3. Study Population

#### **5.3.1.** Target Patient Population

Patients who seek non-invasive fat reduction in the torso region (abdomen, flanks, bra fat, and/or back fat) will be recruited for this study.

#### 5.3.2. Subject Eligibility

To be included in the study, potential subjects must meet all of the inclusion criteria and none of the exclusion criteria listed below.

#### **Inclusion Criteria**

- a) Subject (healthy volunteer) has read and signed the study written informed consent form.
- b) Male or female  $\geq 22$  years and  $\leq 65$  years of age.
- c) Subject has clearly visible fat in one or more areas on the torso (abdomen, flank, back fat, bra fat), which in the investigator's opinion, may benefit from the treatment.
- d) Subject has not had weight change exceeding 5% of body weight in the preceding month.
- e) Subject agrees to maintain his/her weight (i.e., within 5%) by not making any major changes in their diet or exercise routine during the study.
- f) Subject has a BMI  $\leq$  30 as determined at screening.
- g) Subject agrees to have photographs taken of the treatment area(s) during the scheduled time periods.

#### **Exclusion Criteria**

- a) Subject has had a recent surgical procedure in the area of intended treatment.
- b) Subject has had an invasive fat reduction procedure (e.g., liposuction, mesotherapy) in the area of intended treatment.
- c) Subject has had a non-invasive fat reduction and/or body contouring procedure in the area of intended treatment within the past 12 months.
- d) Subject needs to administer or has a known history of subcutaneous injections into the area of intended treatment (e.g., heparin, insulin) within the past month.
- e) Subject has a known history of cryoglobulinemia, paroxysmal cold hemoglobinuria, or cold agglutinin disease.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

f) Subject has a known sensitivity to cold, such as cold urticaria, Raynaud's disease, chilblains (pernio), or any known condition with a response to cold exposure that limits blood flow to the skin.

- g) Subject has a history of bleeding disorder or is taking any medication that in the investigator's opinion may increase the subject's risk of bruising.
- h) Subject is taking or has taken diet pills or supplements within the past month.
- i) Subject has any dermatological conditions, such as moderate to excessive skin laxity, or scars in the location of the treatment sites that may interfere with the treatment or evaluation (stretch marks is not an exclusion).
- j) Subject has an active implanted device such as a pacemaker, defibrillator, or drug delivery system
- k) Subject has a history of hernia in the area(s) to be treated.
- 1) Subject is pregnant or intending to become pregnant during the study period (in the next 8 months).
- m)Subject is lactating or has been lactating in the past 6 months.
- n) Subject is unable or unwilling to comply with the study requirements.
- o) Subject is currently enrolled in a clinical study of any unapproved investigational drug or device.
- p) Any other condition or laboratory value that would, in the professional opinion of the investigator, potentially affect the subject's response or the integrity of the data or would pose an unacceptable risk to the subject.

#### 5.3.3. Vulnerable Populations

Children, pregnant women, fetuses, neonates and prisoners are not included in this study.

## 6. Study Conduct and Procedures

#### 6.1. Recruitment

Potential study subjects will be recruited from clinics of participating investigators as well as through local advertising. Any study-related advertisements will be approved by the governing IRB/EC prior to use.

## 6.2. Informed Consent

Subjects will be recruited from the Investigator's clinical practice and via IRB/EC approved advertising. Once the patient's potential eligibility has been

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

determined, the Investigator or designee trained to the protocol will explain the nature and scope of the study, risks and benefits of participation, answer questions for the subject, and invite the subject to participate. The study will be explained in lay terms. If the patient agrees to participate, the IRB/EC-approved informed consent will be signed and dated by the patient and the Investigator or designee. A copy of the signed and dated informed consent will be provided to the study subject.

#### 6.3. Screening Procedures

After the informed consent is signed, participants will be screened for eligibility. Each participant will be interviewed to determine that all selection criteria are met. The Investigator or designee shall complete a medical history and examine the participant to confirm eligibility for the study. The following activities will be performed at the screening visit:

- 1. Obtain height and weight.
- 2. Calculate BMI. BMI is calculated by multiplying subject weight (in pounds) by 703 divided by the square of the subject's height in inches.
- 3. Assess for any medical conditions that would lead to exclusion of a subject from the study.
- 4. Visually assess and palpate the intended treatment area to determine if it is appropriate for treatment.
- 5. A tissue draw assessment on the treatment sites may be performed to verify the potential subject is a good candidate for CoolSculpting in the torso region such that a minimum of eight cooling cycles can be administered.
- 6. Document medication use, Fitzpatrick Skin Type, and ethnicity.
- 7. Schedule pre-treatment photo visit (to be completed up to 30 days prior to treatment).
- 8. All female subjects of childbearing potential will be asked to take a pregnancy test (urine) prior to being treated. If the subject is pregnant, she will be excluded from participation.

Female participants of childbearing potential will be advised to avoid becoming pregnant during the course of the study by using a medically accepted form of contraception if they are sexually active. If the participant becomes pregnant during the course of the study, she will not be treated subsequently with the study

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

device or be required to have follow-up photographs and ultrasounds taken. Female participants of childbearing potential will be assessed for the start date of their last menstrual cycle.

All participants will be asked to maintain their weight by not making any major changes to their diet or exercise routine during the study. Participants who do not maintain their weight within 5% of their baseline body weight will continue in the study but will be excluded from the effectiveness analyses.

Participants who meet all of the inclusion criteria and none of the exclusion criteria shall be eligible to participate in the study and the first treatment will be scheduled.



Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### 6.6. Treatment Procedures

#### 6.6.1. Treatment Visit #1; Required; Day 0

#### **Prior to CoolSculpting Treatment**

- 1. Review inclusion and exclusion criteria.
- 2. Repeat pregnancy test for female subjects of childbearing potential (urine). Exclude subject from participation if the results are positive.
- 3. If the subjects meet all of the inclusion criteria and none of the exclusion criteria, then proceed with the study treatment.
- 4. Obtain weight
- 5. Obtain baseline photographs of the torso using standardized setup and settings. Alternatively, the baseline photographs may be collected at screening visit.
- 6. Obtain 3-D images.
- 7. Use template to mark the treatment area on each torso area intended for treatment. After marking:
  - a. Insert one geltrap into each slot on back of applicator cup.
  - c. Clean the treatment area with an alcohol wipe.
  - d. Clean the treatment area using a pre-treatment skin wipe.
  - e. Apply CoolAdhesive GelPad on the treatment area per manufacturer's instructions for use.



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



#### 6.6.2. Treatment Visit #2; Required; 6 Weeks (± 1 week)

- 1. Review Inclusion and Exclusion criteria.
- 2. Obtain weight.
- 3. Repeat pregnancy test for female subjects of childbearing potential (urine). Exclude subject from participation if the results are positive.
- 4. Clinical assessment of the treatment area for any epidermal, dermal and subcutaneous findings (e.g., erythema, bruising, swelling, pigment changes) as well as alterations in sensation (e.g., numbness, tingling).
- 5. Assessment of any adverse events.
- 6. Subject feedback via a questionnaire.
- 7. Photography of torso region using the same standardized setup and settings as the pre-treatment photographs (optional).
- 8. Obtain 3-Dimensional images (optional).

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

9. Obtain ultrasound images of the treated area. Ultrasound will be performed by Sponsor staff. (Optional)

10. Perform treatment as described in Section 6.6.1. A minimum of eight treatment cycles will be performed in the study.

## 6.7. Follow-up Procedures

## 6.7.1. One-Week Phone Follow-Up (post-each treatment); Required: 7 Days (± 3 days)

Subjects will be contacted (via phone call or email) one week after Treatment Visit #1 and Treatment Visit #2 to:

- 1. Obtain information regarding the condition of the treatment area
- 2. Obtain subject pain score
- 3. Assess for adverse events

If there is evidence that an adverse event may have occurred, the subject may be asked to come in for a visit so an appropriate evaluation can be performed.



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

## 6.7.3. Twelve-Week Final Follow-up; Required (Day 90 +/- 14 days post-treatment)

The following evaluations will be performed at the 12-week final post-treatment follow-up visit:

- 1. Obtain weight.
- 2. Clinical assessment of the treatment regions for any epidermal, dermal and subcutaneous findings (e.g., erythema, bruising, swelling, pigment changes) as well as alterations in sensation (e.g., numbness, tingling).
- 3. Assessment of any adverse events.
- 4. Subject feedback via questionnaire.
- 5. Standardized and 3D photography of the torso using the same standardized setup and settings as the pre-treatment photographs.
- 6. Obtain ultrasound images of the treated area. Ultrasound will be performed by Sponsor staff. (Optional)

#### 6.7.4. Optional Follow-Up Evaluations (up to 2 within study period)

The full evaluation is not required at optional follow-up visits; the extent of the assessment will be at the discretion of the investigator.

Study activities and events are summarized in **Table 1**, Study Schedule.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

**Table 2. Study Schedule** 

| Study Task | Screening<br>visit<br>(< 1 hr) | Photo Visit<br>(< 1 hr) | Treatment<br>#1<br>( = 4 hrs)</th <th>Treatment<br/>#2<br/>(<!--= 4 hrs)</th--><th>1-Week<br/>Phone<br/>F/U†</th><th>4-Week<br/>F/U Visit†</th><th>12-Week<br/>F/U Visit</th><th>Optional<br/>F/U<br/>Visit**</th></th> | Treatment<br>#2<br>( = 4 hrs)</th <th>1-Week<br/>Phone<br/>F/U†</th> <th>4-Week<br/>F/U Visit†</th> <th>12-Week<br/>F/U Visit</th> <th>Optional<br/>F/U<br/>Visit**</th> | 1-Week<br>Phone<br>F/U† | 4-Week<br>F/U Visit† | 12-Week<br>F/U Visit | Optional<br>F/U<br>Visit** |
|---|---|---|---|---|---|---|---|---|
| | Day -60 to 0 | Day-30 to 1 | Week 1 | Week 6 | Weeks | 30 days | 90 days | Open |
| | | | | | 2 and 7 | (± 7 d) | (+/- 14 d) | |
| Informed Consent | X | | | | | | | |
| Eligibility Criteria | Х | | Х | Χ | | | | |
| Pregnancy Test | Х | | Х | Х | | | | |
| Medical History | Х | | | | | | | |
| Height | Х | | | | | | | |
| Weight | Х | Х | Х | Χ | | Х | Χ | |
| Photography-2D & 3D<br>Baseline & 3 month<br>required | | X* | | Х* | | X* | X* | |
| Ultrasound (optional) | | X* | | Х* | | Х* | Х* | |
| Satisfaction Questionnaire | | | | Χ | | Х | Χ | |
| CoolSculpting Treatment | | | Х | Χ | | | | |
| Pain Assessment | | | Х | Х | Х | Х | Χ | |
| AE Assessment | Х | Х | Х | Х | Х | Х | Χ | Х |

X\* indicates procedures which may be performed by staff of the Sponsor

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

<sup>\*\*</sup> Investigator discretion as to timing and extent of follow-up assessment for optional visits.

 $<sup>\</sup>dagger$  Follow-up after each treatment

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



## 7. Statistical Methodology and Analyses

## 7.1. Primary Endpoints

The primary endpoints of the study are defined as follows:

- Safety Endpoint: The frequency of device-related adverse events (AEs) including device-related serious adverse events (SAEs) will be summarized.
- Efficacy Endpoint: The primary effectiveness endpoint is the correct identification of pre-treatment vs. 12-Week post-treatment images by at least two out of three blinded, independent reviewers. Success is defined as at least 70% correct identification of the pre-treatment images.

#### 7.2. Statistical Methods: Overall Plan

Data will be summarized based on the nature of the data. Dichotomous (e.g., gender, independent photographic review) and ordinal (e.g., Fitzpatrick Skin type) data will be tabulated by category. The mean, standard deviation, maximum, and minimum will be tabulated for continuous data (e.g., age, fat thickness). The significance level will be two-sided 0.05 for all statistical tests.

## 7.3. Analysis Cohorts

#### 7.3.1. Safety Cohort

This cohort will consist of all the treated participants with safety evaluation after the treatment. This cohort should be identical to the As Treated (AT) cohort. The safety data analyses will be performed based on the Safety Cohort.

#### 7.3.2. Effectiveness Cohorts

Two groups of subjects will be identified for the analysis of effectiveness endpoints: Per Protocol Cohort and the As Treated Cohort. All analyses of

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

effectiveness will be performed on each cohort of subjects. However, study success will be based on the Per Protocol Cohort of subjects.

#### **Per-protocol Cohort (PP):**

The Per-protocol Population will consist of all the treated subjects (completing 2 treatment sessions with at least 8 total cycles) followed through to the final post-treatment visit and with weight change of no more than  $\pm 5\%$  at the time the final post-treatment visit images are taken. Since a weight change of more than 5 percent will affect the images, the primary efficacy analysis will be performed based on this study population.

#### **As-Treated Cohort (AT):**

This cohort consists of all treated participants regardless of whether they become pregnant or undergo weight change during the study.

#### 7.3.3. Endpoint Analysis

#### **Primary Safety Endpoint**

The primary safety endpoint will be the frequency of device-related adverse events (AEs) including device-related serious adverse events (SAEs). The number and percentage of subjects experiencing each AE will be descriptively summarized. Adverse events and SAEs will be presented as summary tables showing the frequency and type of events.

#### **Primary Efficacy Endpoint:**

The primary efficacy endpoint is the correct identification of pre-treatment vs 12-week post-treatment images. Since weight change will affect the image, the analysis will be based on the evaluation of the PP population, i.e. treated subjects followed for 12 weeks who did not became pregnant, and with weight change of no more than  $\pm 5\%$  at the 12-week visit. Success will be defined as at least 70% correct identification of the pre-treatment images.

#### 7.3.4. Missing Data Handling:

In general, no imputation for missing data will be made. Data will be analyzed "as-is" where subjects with missing data not being included in the analysis.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### 7.3.5. **Data Pooling:**

Data are assumed to be poolable across sites due to: 1) use of the same study protocol, 2) equivalent training of all sites in the study protocol and use of the investigational device, 3) use of the same CRF at each site, and 4) use of Independent Evaluator(s).



#### 8. Adverse Events

Adverse events (AE) will be assessed continuously throughout the study. An AE is defined in accordance with ISO 14155 as any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in study participants, users, or other persons temporally associated with the use of study treatment, whether or not considered related to the study treatment. <sup>2</sup>

Disease signs and symptoms that existed prior to the study treatment are not considered AEs unless the condition recurs after the patient has recovered from the pre-existing condition or the condition worsens in intensity or frequency during the study.

AEs will be monitored throughout the study beginning with signing of informed consent. At each post-baseline visit, the investigator will begin querying for AEs by asking each patient a general, non-directed question such as "Have you had any changes to your condition since your last visit?" Previous AEs and changes in therapy/concomitant medications are to be updated. Directed questioning and examination will then be done as

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001

(OneV-83717 Ver 2.0)

<sup>&</sup>lt;sup>2</sup> Clinical Investigation of medical devices for human subjects – Good Clinical Practice (ISO 14155:2011)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

appropriate. All reportable AEs and clinically significant abnormal laboratory findings will be documented on the appropriate CRF.

Adverse events will be reported by the participant (or, when appropriate, by a caregiver, surrogate, or the participant's legally authorized representative). The investigator and any designees are responsible for detecting, collecting and recording events that meet the definition of an AE or SAE and remain responsible for following up AEs that are serious, considered related to the study treatment or study procedures, or that caused the participant to discontinue the study until the event has resolved or until 30 days after the completion of the study.

## 8.1. Adverse Device Effect (ADE)

Any sign, symptom, or disease in a study subject that occurs during the course of a clinical trial that is determined by the Investigator to have a causal relationship or possible causal relationship with the device under investigation. This definition includes any AE s resulting from insufficient or inadequate instructions for use, deployment, implantation, installation, or operation, or any malfunction of the investigational medical device as well as any event resulting from use error (per ISO 62366) or from intentional misuse of the investigational medical device.

#### 8.1.1. Serious Adverse Device Effect (SADE)

A serious adverse device effect (SADE) is defined in accordance with ISO 14155 as "an adverse device effect that has resulted in any of the consequences characteristic of a serious adverse event."

#### 8.1.2. Unanticipated Serious Adverse Device Effect (USADE)

An unanticipated serious adverse device effect (USADE) is defined in accordance with ISO 14155 as "any serious adverse device effect which by its nature, incidence, severity, or outcome has not been identified in the current version of the risk analysis report." The investigator is to consult the IFU for anticipated risks or anticipated AEs.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### 8.1.3. Serious Adverse Event (SAE)

An SAE is defined in accordance with ISO 14155 as an AE that:

- 1. Led to death
- 2. Led to serious deterioration in the health of the patient, that either resulted in:
  - a. a life-threatening illness or injury, or
  - b. a permanent impairment of a body structure or a body function, or
  - c. inpatient or prolonged hospitalization, or
  - d. medical or surgical intervention to prevent lifethreatening illness or injury or permanent impairment to a body structure or a body function, or
  - e. led to fetal distress, fetal death or a congenital abnormality or birth defect

NOTE: Planned hospitalization for a pre-existing condition, or a procedure required by the protocol, without serious deterioration in health, is not considered an SAE.

#### 8.1.4. Time Period and Frequency for Collecting AE and SAE Information

All AEs and SAEs from the signing of the Informed Consent Form (ICF) until the last follow-up visit will be collected at the time points specified in the schedule of activities, and as observed or reported spontaneously by study participants.

Medical occurrences that begin after signing of informed consent and before administration of study treatment will be recorded as an AE on the appropriate CRF.

All SAEs will be recorded and reported to the Sponsor or designee within 24 hours of learning about the report. All non-serious AEs related to the devices used in the study, as well as Device Complaints, will be reported to the Sponsor within 7 working days. The investigator will submit any updates on these events to the Sponsor within 24 hours of it being available.

Investigators are not obligated to actively seek AE or SAE in former study participants. However, if the investigator learns of any SAE, including a death, at any time after a participant has completed the final visit of the

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

study, and he/she considers the event to be reasonably related to the study treatment or study participation, the investigator must promptly report the event to the Sponsor.

#### 8.1.5. Method of Detecting AEs and SAEs

Care will be taken not to introduce bias when detecting AEs and/or SAEs. Open-ended and non-leading verbal questioning of the participant is the preferred method to inquire about possible AEs.

#### 8.1.6. Follow-up of AEs and SAEs

After the initial AE/SAE report, the investigator is required to proactively follow each participant at subsequent visits/contacts. All SAEs will be followed until resolution, stabilization, the event is otherwise explained, or the participant is lost to follow-up or until 30 days after completion of the study.

The investigator is obligated to perform or arrange for the conduct of supplemental measurements and/or evaluations as medically indicated or as requested by the Sponsor to elucidate the nature and/or causality of the AE or SAE as fully as possible. This may include additional laboratory tests or investigations, histopathological examinations, or consultation with other health care professionals.

New or updated information will be recorded in the originally completed CRF.

The investigator will submit any updated SAE data to the Sponsor within 24 hours of receipt of the information.

#### 8.1.7. Reportable Incidents

Serious adverse events (SAEs and SADEs) as well as unanticipated adverse device effects (UADEs) must be reported within 24 hours of knowledge of the event to the Sponsor.

All adverse events observed by the investigator or reported by the subject will be recorded on the appropriate CRF, irrespective of the relationship to the investigational device used in the study. Medically significant adverse events will be followed until resolved or considered stable. For each event, the investigator will record a description, dates of onset and resolution, severity, and relationship to the investigational device. The investigator may

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

be required to provide follow-up information as-needed to fulfill requirements for regulatory reporting.

Any adverse event that results in withdrawal from the study must be reported to the Sponsor after the decision to withdraw the subject is made.

Any death occurring during the study must be reported to the Sponsor within 24 hours.

If an event is classified as an SADE or a UADE, the Sponsor will determine if there is an unreasonable risk to the patients within the study. In the event a UADE is reported during this study, it will be reported to the IRB and to the regulatory agencies as appropriate according to the relevant standard operating procedures and law of the country where the trial is performed.

#### 8.1.8. Assessment of Severity

Severity of adverse events will be determined using the following scale:

- <u>Mild</u>: Event that is easily tolerated and may require only minimal treatment or therapeutic intervention. The event does not generally interfere with usual activities of daily living.
- <u>Moderate</u>: Events that interfere with usual activities of daily living, causing discomfort but poses no significant or permanent risk of harm to the research participant. It is usually alleviated with additional specific therapeutic intervention.
- <u>Severe</u>: Event that is incapacitating, with inability to work and do the usual activities of daily living, or significantly affects clinical status. This may require intensive therapeutic intervention.

#### 8.1.9. Assessment of Relatedness

- The investigator is obligated to assess the relationship between study treatment and each occurrence of each AE/SAE.
- A *reasonable possibility* of a relationship conveys that there are facts, evidence, and/or arguments to suggest a causal relationship, rather than a relationship cannot be ruled out.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

• The investigator will use clinical judgment to determine the relatedness.

- Alternative causes, such as underlying disease(s), concomitant therapy, and other risk factors, as well as the temporal relationship of the event to study treatment administration will be considered and investigated.
- The investigator will also consult the investigator's brochure and/or product information, for marketed products, in his/her assessment.
- For each AE/SAE, the investigator must document in the medical notes that he/she has reviewed the AE/SAE and has provided an assessment of relatedness.
- For each AE/SAE, there are 4 levels of relatedness, as follows:
  - Not related
  - Possible
  - Probable
  - Definite relationship

There may be situations in which an SAE has occurred and the investigator has minimal information to include in the initial report to the Sponsor. However, it is very important that the investigator always make an assessment of relatedness for every event before the initial transmission of the SAE data to the Sponsor.

- The investigator may change his/her opinion of relatedness in light of follow-up information and send an SAE follow-up report with the updated relatedness assessment.
- The relatedness assessment is one of the criteria used when determining regulatory reporting requirements.

The investigator will determine the relationship of each adverse event to the study device using the question: "Is there a reasonable possibility that the

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

event may be related to treatment with the device? Answer 'yes' or 'no' for each adverse event."

The guideline below should be used to consider relatedness:

For a "not related" assessment, the adverse event:

- May be judged to be due to extraneous causes such as disease or environment or toxic factors
- May be judged to be due to the subject's clinical state or other therapy being administered
- Is not biologically plausible
- Does not reappear or worsen when the investigational device is re-administered
- Does not follow a temporal sequence from treatment with the investigational device,

For an assessment of relatedness (including, probable and possible assessments) there is a reasonable possibility that the event may have been caused by the investigational device, the adverse event:

- Follows a temporal sequence from treatment with the device.
- Is a known response to the device based on clinical or nonclinical data
- Could not be explained by the known characteristics of the subject's clinical state, environmental or toxic factors, or other therapy administered
- Disappears or decreases upon cessation of the use of the device.
- Reappears or worsens when the device is readministered.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### 8.1.10. Serious Adverse Event Reporting Procedures

All serious adverse events must be reported to the Sponsor within one (1) working day of discovery or notification of the event and according to IEC/IRB requirements and the institution at which the study is conducted, if applicable. Serious adverse event information and any follow-up information will be recorded on a Serious Adverse Event Form and transmitted to the Sponsor using the contact information provided by the Sponsor. Note that for each device used in this study, a separate SAE form and contact information will be used. The Sponsor is responsible for evaluating and reporting any serious adverse event and unexpected serious adverse reactions in accordance with all applicable laws and standards.

#### **Reportable Incidents**

Serious adverse events (SAEs) and unanticipated adverse device effects (UADEs) must be recorded and reported to the Sponsor or designee within 24 hours of knowledge of the event to the Sponsor:

ZELTIQ Aesthetics, an Allergan affiliate 4410 Rosewood Dr.
Pleasanton, CA 94588
PH:

A full reporting of the event shall be provided within 10 working days of the event. The Sponsor is then responsible for notifying the IRB, as required.

Other adverse events, deemed by the Investigator to be non-serious, should be provided to the Sponsor as soon as possible and not later than 1 week after knowledge of the event. This will be forwarded to the Product Surveillance team within 24 hours of receipt by the Sponsor Contact.

Additional information obtained by the Clinical Site regarding any adverse event, both serious and non-serious, will be reported to the Sponsor within 24 hours of awareness.

#### **Safety Monitoring Considerations**

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

If an adverse event occurs that in the judgment of the investigator represents a potential risk for new subjects, the investigator will contact the Sponsor within 1 working day after becoming aware of the event.

A full reporting of the event shall be provided within 10 working days of the event. The Sponsor is then responsible for notifying the IRB/EC, as required.

#### 8.1.11. Pregnancy

- Details of all pregnancies in female participants will be collected after the start of study treatment through the duration of the pregnancy.
- If a pregnancy is reported, the investigator should inform the Sponsor within 24 hours of learning of the pregnancy.
- If a female of childbearing potential becomes pregnant during the study, the investigator should notify the participant's physician that the participant may have been treated with the investigational device and exit the participant from the study.
- Abnormal pregnancy outcomes (e.g., spontaneous abortion, fetal death, stillbirth, congenital anomalies, ectopic pregnancy) are considered SAEs.

## 9. Device Tracking

The Sponsor will send the Investigator investigational devices. The Investigator must house study devices in an appropriate, secure location.

The Sponsor will track sending and receiving of devices to/from the Investigator. The Investigator must track receipt and final disposition of the devices, and maintain accurate records of the use of the device on each study subject.

In addition, for IDE studies, the Investigator must maintain records of receipt, use and disposition of all devices on a device accountability log which will be monitored by the Sponsor and a copy collected at the end of the study. An accurate record of the date the device was used on each subject must be available for inspection at any time.

## 9.1. Device Packaging and Labeling

Clinical study devices will be packaged and labeled according to the country's regulatory requirements.
Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

The study device or its immediate package, will be labeled per the requirements of 21CFR 812.5(a).

## 10. Device Deficiencies and Malfunctions

A device deficiency is defined in accordance with ISO 14155 as "inadequacy of a medical device with respect to its identity, quality, durability, reliability, safety, or performance." Device deficiencies include malfunctions, use errors, and inadequate labeling.

If a device deficiency occurs, the investigator will notify the Sponsor. Device deficiencies shall be documented throughout the study and appropriately managed and reported to regulatory authorities and IRBs as required by national regulations.

# 11. Ethical and Regulatory Considerations

## 11.1. Compliance with Good Clinical Practice

This study will be conducted in compliance with the principles of the Declaration of Helsinki, with the current Good Clinical Practice (GCP) guidelines and with other applicable regulations. The Investigator and all study staff will conduct the study in compliance with this protocol. Voluntary informed consent will be given by every subject prior to the initiation of any study-related procedures. The rights, safety and well-being of the study subjects are the most important considerations and prevail over the interests of science and society. All personnel involved in the conduct of this study must be qualified by education, training and experience to perform their assigned responsibilities.

# 11.2. Institutional Review Board (IRB) and Informed Consent

Before study initiation, the Investigator must have written and dated approval from the IRB/EC for the protocol, consent form, subject recruitment materials/process (e.g., advertisements), and any other written information to be provided to subjects. The Investigator should also provide the IRB/EC with a copy of the product labeling, information to be provided to subjects and any updates. The Investigator will submit documentation of the IRB/EC approval to the Sponsor. Copies of all correspondence with the IRB/EC regarding this study must be sent to the Sponsor.

The IRB/EC-approved consent form must include all elements required by FDA, state, and local regulations, and may include appropriate additional elements.

The Investigator/designee will explain the study to each potential subject and the subject must indicate voluntary consent by signing and dating the approved informed consent form. The Investigator must provide the subject with a copy of the consent form in a

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

language the subject understands. The Investigator will maintain documentation that informed consent was obtained prior to the initiation of any study-specific procedures.

Withdrawal of IRB/EC approval of the Investigator's part in the investigation must be reported to the Sponsor within 5 working days.

#### 11.3. Protocol Adherence

The study investigators are responsible for performing the study in compliance with the protocol. Non-adherence to the protocol is to be classified as a protocol violation, protocol deviation, as defined below.

#### **Protocol Violation**

Non-adherence to the protocol that may result in significant additional risk to the participant (e.g., enrollment of a participant who does not meet the study criteria). Or, non-adherence to Good Clinical Practices (GCP) that may impact patient safety (e.g., failure to obtain proper consent prior to performing study procedures). Violations should be reported to the study Sponsor and the IRB within 5 working days if they occur.

#### **Protocol Deviation**

Non-adherence to study procedures which does not result in additional risk to the participant (e.g., participant missed visit). Protocol deviations are not required to be reported to the IRB; however, they must be recorded and addressed on the study case report forms and may be reported and reviewed in conjunction with the progress report as part of the annual review process.

#### **Protocol Waivers**

Waivers, exceptions or any intentional deviation from the approved protocol are not permitted in the study.

#### 11.4. Protocol Amendments

Amendments to the study protocol can be made only by the study Sponsor. A revised protocol can be put into place only after governing IRB/EC approval. All administrative letters must be submitted to the IRB/EC for their information.

New or altered consent forms required by the IRB due to a protocol change must be used for any subsequent subject enrollment and when the IRB requires, signed by subjects currently enrolled in the study.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

# 12. Study Management and Quality Control

### 12.1. Study Data Collection

Zeltiq will supply Case Report Forms (CRFs) to all participating sites for this study.

A CRF is required and will be completed for each included subject. The Investigator has ultimate responsibility for the collection and reporting of all data entered on the CRFs and any other data collection forms (source documents) and ensuring that they are accurate, authentic/original, attributable, complete, consistent, legible, timely (contemporaneous), enduring and available when required. The CRFs must be signed by the Investigator to attest that the data contained therein are true.

### Paper Based CRFs

Demographic, Screening (Inclusion/Exclusion), Treatment, Follow Up, Adverse Event, Protocol Deviation, and Study Termination Data will be recorded on paper Case Report Forms (CRFs) developed by the Sponsor. Completed CRFs will be monitored by the Sponsor or a designee at defined intervals and the original CRFs will be collected. Copies will remain filed at the investigational sites. The data will then be reviewed by the Sponsor and entered into a study database. Data queries will be issued as necessary to clarify discrepancies.

## 12.2. Data Management

Data management activities will be performed in accordance with internal Zeltiq SOPs for handling data in non-significant risk studies conducted under abbreviated IDE requirements.

### 12.2.1. Data Receipt and Data Entry

The monitor will collect clinical study related documents including Case Report Forms (CRFs), Data Clarification Forms (DCFs), and any other clinical documents from clinical sites and transmit the documents to the Sponsor as appropriate.

# 12.3. Confidentiality

All information and data concerning study participants will be considered confidential, and handled in compliance with all applicable regulations including the requirements of the Health Insurance Portability and Accountability Act (HIPAA) of 1996.

ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

The investigator is responsible for ensuring the confidentiality of subjects throughout the trial. A unique identification code will be assigned to each subject participating in this trial. Any data that may be published in abstracts, scientific journals, or presented at medical meetings will reference a unique subject code and will not reveal the subject's identity.

Only authorized site staff, the study Sponsor or the Sponsor's designee, IRB/EC or regulatory authorities will have access to these confidential files. All data used in the analysis, reporting and publication of this clinical trial will be maintained without identifiable reference to the participant. Any data that may be published in abstracts, scientific journals, or presented at medical meetings will reference a unique participant code and will not reveal the participant's identity.

### 12.4. Quality Assurance Audits

Sponsor representatives or designees may conduct site quality assurance (QA) audits during the study. The Investigator must agree to provide the auditor with direct access to all relevant documents and discuss any findings with the auditor.

In the event of an inspection by the FDA or other regulatory authorities, the Investigator must give the inspector direct access to relevant documents and to discuss any findings with the inspector. The Investigator must notify Zeltiq in the event of a FDA site audit.

# 12.5. Investigator Responsibilities

#### 12.5.1. General Responsibilities

Investigators are responsible for ensuring the investigation is conducted according to all signed agreements, the Protocol, and applicable FDA regulations. The investigator must protect the rights, safety, privacy and welfare of the participants under the Investigator's care. Investigators will assume overall responsibility and accountability for study site staff and for the clinical data obtained during the study. The investigator assumes all responsibilities per applicable regulations, including but not limited to:

**IRB approval**: The investigator may not begin the study until the FDA and the governing institutional review board (IRB) provide written approval of the study protocol and consent form. The investigator is also responsible for fulfilling any conditions of approval imposed by the IRB.

**Informed Consent**: The investigator must ensure that informed consent is obtained from each prospective study participant in accordance with 21 CFR

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

Part 50 and that the study is not commenced until FDA and IRB approvals have been obtained.

**Financial Disclosure:** Investigators shall provide financial disclosure according to federal regulations.

**Study Coordinator:** To assure proper execution of the study protocol, each investigator must identify a study coordinator for the site who will work with and under the authority of the investigator to assure that study requirements are fulfilled as appropriate.

#### 12.5.2. Investigator Records

The investigator and study staff must maintain accurate, complete, and current records relating to the conduct of the investigation. Records must be retained for a period of two years following (1) the date the investigation was completed or terminated, or (2) the records are no longer required to support a regulatory submission or completion of a product development protocol, whichever is longer. Participating investigators shall maintain the following:

- All correspondence with the Sponsor, another investigator, the IRB, a monitor, or the FDA
- Records of all persons authorized to conduct the study (e.g. Delegation of Duties/Signature Authorization, CV)
- Records of receipt, use or disposition of the device
- Informed Consent documentation for all enrolled participants
- Records of each participant's case history, including study-required Case Report Forms and source documentation (e.g. physician notes, lab reports, study worksheets, clinic charts)
- All relevant observations of adverse device effects
- Records of any protocol deviations
- The condition of each participant upon entering and during the course of the investigation and any relevant medical history and results of any diagnostic tests
- Record of each participant's exposure to the device, including the date and time of use

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

Protocol with all amendments

- Current IRB approved informed consent and all previously approved versions
- Signed Investigator Agreement
- Investigators will be responsible for the accurate and timely completion of CRFs during the trial.

These records must be available and suitable for inspection at any time by Sponsor representatives (monitor), the reviewing IRB, or FDA. The Investigator will supply access to study-related medical records, original laboratory data, and other records and data as they relate to the trial. The investigator will ensure that both he/she and his/her study staff have adequate time and resources to devote to the study, including study enrollment, participant evaluations, study documentation and site monitoring.

### 12.5.3. Investigator Reports

The investigator is responsible for preparation and submission of the following reports:

- Report of any unanticipated adverse device effects shall be submitted to the Sponsor within 24 hours and no later than 10 working days after the Investigator first learns of the effect
- Withdrawal of IRB approval of the investigator's part in the investigation shall be reported to the Sponsor within 5 working days
- Progress reports on the investigation to the sponsor, the monitor, and the reviewing IRB annually. Alternatively, the Sponsor may prepare the report.
- Deviations from the protocol shall be reported to the Sponsor and the IRB
- Failure to obtain informed consent prior to use of a device in a participant shall be reported to the Sponsor and IRB within 5 working days after the use occurs
- A final report shall be submitted to the Sponsor and IRB within 3 months after termination or completion of the investigation, or the investigator's part of the investigation.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

## 12.6. Sponsor Responsibilities

#### **12.6.1.** General Responsibilities:

As the Sponsor, ZELTIQ Aesthetics assumes overall responsibility for the conduct of the study including assurance that the study satisfies applicable regulatory requirements. ZELTIQ Aesthetics assumes all responsibilities per applicable regulations, and shall:

**IRB approval:** Ensure IRB approval for the investigation. No IDE application is necessary for this study.

**Investigators**: Select investigators qualified by training and experience, and providing them with the information they need to conduct the study properly. Obtain a signed Investigator Agreement from each participating investigator. Study sites will be evaluated to ensure that they have an adequate participant base and can provide sufficient staff and documentation support to conduct the study properly.

**Monitoring**: Select monitors qualified by training and experience and ensure proper monitoring of the study.

**Data Management and analysis:** Ensure data collection, verification, analysis, records storage, etc. Sponsor will assist with presentation(s) and/or publication(s).

**Essential Document Records:** Maintain all Essential Documents pertaining to the study per ISO 14155:2011. Records must be retained for a period of two years following (1) the date the investigation was completed or terminated, or (2) the records are no longer required to support a regulatory submission or completion of a product development protocol, whichever is longer.

**Study Training:** To ensure uniform data collection and protocol compliance, Sponsor personnel will provide an educational session to study site personnel which will cover the Protocol, techniques for the identification of eligible participants, data collection and form completion, and the device directions for use. The investigator and study staff will be trained on the study device and protocol, applicable regulations and requirements, and expectations of

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

the study, enrollment expectations, participant selection, informed consent, required clinical data and record keeping, etc.

**Device Use:** Representatives of the Sponsor will train investigators in use of the study device.

#### 12.6.2. Site Monitoring

The Sponsor will ensure that qualified clinical monitors are available to monitor and oversee the conduct of the trial and that monitoring is performed in accordance with the Sponsor's approved procedures or third-party procedures approved by the Sponsor.

The clinical monitors will evaluate compliance with the protocol and applicable regulations, any specific recommendations made by the site's IRB and the signed Investigator Agreement.

#### **Monitoring Visits**

On-site monitoring visits will assess the progress of the clinical study and identify any concerns that result from device performance or review of the investigator's study records, study management documents, and informed consent documents.

Monitoring will ensure continued protocol compliance, accurate data reporting, and adequate accounting of shipments of study devices.

The study design includes two treatment visits with the final visit occurring 3 months post-final treatment. A monitoring visit will occur after the treatment visits are completed, and at least one additional monitoring visit will occur at each site prior to, or in conjunction with, study closeout.

In the event that monitoring identifies serious and/or persistent noncompliance of an investigator, the issue will be escalated to Zeltiq Clinical management.

During monitoring visits, the monitor will compare participant records and other supporting documents with reports at the site to determine that:

• The facilities used by the investigation continue to be acceptable for the purposes of the clinical study

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

 Informed consent was properly obtained and documented for all enrolled study participants

- The protocol is being followed, and only eligible participants are being enrolled into the study
- Deviations to the Protocol have been reported to ZELTIQ and the IRB, as appropriate
- Adverse events are promptly being reported
- Device accountability is being maintained
- Information recorded in the case report forms and study reports are accurate, complete, legible and consistent with source documentation
- Participants failing to complete the clinical study and the reason for failure are recorded
- Missed follow-up visits are noted in the study documentation

Clinical monitors will provide feedback to the site regarding protocol or study compliance. If monitoring reveals significant Investigator noncompliance with the study agreements, protocol, applicable regulations, IRB approval conditions, the monitor will notify Sponsor Clinical Management. Action will be taken to secure compliance, and if further compliance problems persist, or the issue is deemed serious (i.e. endangering patient welfare or safety), the site may be removed from the study and/or the investigator disqualified from future studies.

### **Study Site Closeout**

At the close of the study at an investigational site, the monitor will make a final on-site visit to ensure that all case report forms have been monitored and retrieved and that the investigator's files are accurate and complete. The monitor will ensure that all investigational devices and study supplies are accounted for, and provide for appropriate disposition of any remaining supplies. The monitor will review record retention requirements with the investigator and any remaining investigator obligations are reviewed and ensure that all applicable requirements are met for the study. The monitor will prepare a report of the site closeout visit. The closeout visit may be combined with a final monitoring visit.

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System

#### 12.6.3. Final Report

A final report will be prepared at the conclusion of the trial. Copies of the final report will be provided to each investigator and to the respective IRBs.

#### 12.6.4. Trial Registration

When appropriate, prior to study initiation, the trial will be registered on a publicly accessible study database such as clinicaltrials.gov.

# 13. Data Ownership

ZELTIQ Aesthetics, the study Sponsor, retains ownership of all data generated in this study, and controls the use of the data for purposes of regulatory submissions to the US and/or other governments. Investigator(s) and institution(s) (which shall include their employees, agents, and representatives) may not issue or disseminate any press release or statement, nor initiate any communication of information regarding this study (written or oral) to the communications media or third parties without the prior written consent of the Sponsor.



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)

Part Number: CS-305578 Revision: 04 

Title: Noninvasive Fat Reduction with the CoolSculpting System



ZELTIQ P/N: CS-305578-04 Protocol Number: ZA20-001 (OneV-83717 Ver 2.0)